CLINICAL TRIAL: NCT03479320
Title: Efficacy of Perioperative Intravenous Lidocaine Infusion on Postoperative Analgesia in Patients Undergoing Oral and Maxillofacial Surgeries Under General Anesthesia
Brief Title: Usefulness of Lidocaine in Oral and Maxillofacial Surgeries Under General Anesthesia for Pain Control After Operation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Vivek Kumar Mahato, Post graduate resident in Department of Oral and Maxillofacial Surgery, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRC/1078/017
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Lidocaine group will receive intravenous bolus 1.5 mg/kg at induction followed by continuous infusion of 2 mg/kg/hr until the completion of surgery
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): They will receive the same volume of 0.9% of normal saline as calculated for the experimental group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Postoperative analgesic effects will be compared between lidocaine and normal saline group
  Arms: Lidocaine group
Drug: Placebo — Postoperative anlagesic requirements will be calculated and compared with experimental group
  Arms: Placebo

SUMMARY:
This will be a randomized double blinded clinical study conducted in patients undergoing oral and maxillofacial surgery under general anesthesia. Lidocaine group will receive intravenous bolus 1.5 mg/kg at induction followed by continuous infusion of 2 mg/kg/hr until the completion of surgery.Normal saline group will receive same amount of intravenous normal saline .The primary outcome will be postoperative pain using the NRS scale during first 24 hours and time to first analgesic request

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-60 years of age
* Patients of ASA (American Society of Anesthesiologists) Class I or Class II (I- healthy with no systemic disease, II- mild systemic disease with no functional limitation) who require oral and maxillofacial surgeries under general anesthesia

Exclusion Criteria:

* Refusal to give consent.
* Hypersensitivity or allergy to the study medication.
* ASA physical status III or more.
* Subjects with known severe hepatic or renal dysfunction or cardiac dysrhythmia or atrioventricular block.
* History of taking opioids or antiarrhythmic drugs within 1 week of surgery.
* History of drug or alcohol abuse
* History of psychiatric disorders.
* Patients requiring emergency surgery.
* Patients unable to comprehend pain assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Postoperative Numeric Rating Scale(NRS) | 24 hours
  Pain at rest and with cough or movement using the NRS scale, which ranges from 0 to 10; where 0 refers to no pain and 10 refers to most severe pain

SECONDARY OUTCOMES:
Total opioid consumption | 24 hours
  Total morphine or morphine equivalent in milligram
Time to first analgesic request | 24 hours
  Time to first analgesic (ketorolac) request (time counted after skin closure)
Side effects | 24 hours
  Number of patients with light headedness, sedation, nausea, vomiting will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Kr Mahato, BDS, Principal Investigator — B.P. Koirala Institute of Health Sciences
Locations (1):
- B. P. Koirala Institute of Health Sciences, Dharān, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahato VK, Dongol A, Acharya P, Yadav AK, Subedi A, Jaisani MR. "Can Perioperative Intravenous Lidocaine Decrease Postoperative Pain After Oral and Maxillofacial Surgeries?": A Randomized Clinical Trial. J Maxillofac Oral Surg. 2024 Oct;23(5):1240-1247. doi: 10.1007/s12663-022-01831-1. Epub 2022 Dec 20. PMID 39376771